CLINICAL TRIAL: NCT02210806
Title: Efficacy, Dose-ranging and Safety Evaluation (A Randomized, Double- or Evaluator-blinded, Active- and Placebo-controlled, Single Dose, Five-arm, Crossover, and Dose-ranging Study of A006 in Adult Asthma Patients)
Brief Title: Albuterol DPI (A006) Clinical Study-B3:Efficacy, Dose-ranging and Safety Evaluation
Acronym: A006-B3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: API-A006-CL-B3
Record Dates: First submitted 2014-08-04; First posted 2014-08-07 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Asthma
Keywords: Asthma; Mild-to-moderate persistent asthma; Mild asthma; Moderate asthma; Persistent asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment T1 (Active Comparator): One inhalation of 110 mcg A006 DPI. Total 110 mcg.
  Interventions: Drug: A006 DPI
- Treatment T2 (Active Comparator): One inhalation of 220 mcg A006 DPI. Total 220 mcg.
  Interventions: Drug: A006 DPI
- Placebo (Placebo Comparator): One inhalation of placebo DPI . Total 0 mcg
  Interventions: Other: Placebo DPI
- Treatment R1 (Active Comparator): One inhalation of Proventil® MDI Total 90 mcg
  Interventions: Drug: Proventil® MDI
- Treatment R2 (Active Comparator): Two inhalations of Proventil® MDI, 180 mcg total
  Interventions: Drug: Proventil® MDI

INTERVENTIONS:
Drug: A006 DPI — Single dose 110 mcg, 1 inhalation
  Other Names: Albuterol; Albuterol DPI
  Arms: Treatment T1
Drug: A006 DPI — Single dose 220 mcg, 1 inhalation
  Other Names: Albuterol; Albuterol DPI
  Arms: Treatment T2
Other: Placebo DPI — Placebo, 1 inhalation
  Other Names: Placebo
  Arms: Placebo
Drug: Proventil® MDI — Single dose 90 mcg, 1 inhalation
  Other Names: Proventil®
  Arms: Treatment R1
Drug: Proventil® MDI — Single dose 90 mcg, 2 inhalations
  Other Names: Proventil®
  Arms: Treatment R2

SUMMARY:
This study evaluates the efficacy, dose-ranging and safety profiles of A006, an Albuterol dry powder inhaler (DPI), in the dose range of 110 to 220 mcg per dose in comparison to a DPI Placebo Control and an Albuterol metered dose inhaler (MDI) Active Control.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety profiles of A006 and to assist in identifying the optimum dose of A006 for future clinical studies. Proventil® HFA MDI, a currently marketed Albuterol MDI product, will be used as an Active Control. The study also employs a Placebo Control DPI, which has the same configuration as the A006 DPI except that it contains no active ingredient.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, male and female adults, 18-55 years of age at Screening
* With mild-to-moderate persistent asthma for at least 6 months prior to Screening, and having used inhaled β-agonist(s) for asthma control
* Demonstrating a Screening Baseline FEV1 at 50.0 - 85.0% of predicted normal
* Demonstrating a ≥ 15.0% Airway Reversibility in FEV1 within 30 min after inhaling 2 actuations of Proventil® MDI (180 mcg) at Screening
* Demonstrating Peak Inspiratory Flow Rate (PIF) within 80-150 L/min (after training), for at least 2 times consecutively with a maximum of 5 attempts
* Demonstrating proficiency in the use of a DPI and an MDI after training
* Females of child-bearing potential must be non-pregnant, non-lactating; both males and females enrolled into the study must agree to practice a clinically acceptable form of birth control (including but not limited to, abstinence, double barrier, etc)
* Having properly consented to participate in the trial

Exclusion Criteria:

* A smoking history of ≥ 5 pack-years, or having smoked within 6 months prior to Screening
* Upper respiratory tract infections or lower respiratory tract infection within 6 weeks, prior to Screening
* Asthma exacerbations that required emergency care or hospitalized treatment, within 4 weeks prior to Screening
* Any current or recent respiratory conditions that, per investigator discretion, might significantly affect pharmacodynamic response to the study drugs, including cystic fibrosis, bronchiectasis, tuberculosis, emphysema, and other significant respiratory diseases besides asthma
* Concurrent clinically significant cardiovascular (e.g. hypertension and tachyarrhythmia and bradyarrhythmia), hematological, renal, neurologic, hepatic, endocrine, psychiatric, malignant, or other illnesses that in the opinion of the investigator could impact on the conduct, safety and evaluation of the study
* Known intolerance or hypersensitivity to any of the ingredients of the study drug DPI or Proventil® HFA MDI (i.e., Albuterol, sulfate, lactose, milk protein, HFA-134a, oleic acid, and ethanol)
* Baseline ECG at Screening or Visit 1 showing any single or multiple premature ventricular contractions (PVC)
* Baseline ECG at Screening or Visit 1 with a confirmed (through performing a second ECG) QTc reading greater than 450ms
* Use of prohibited drugs or failure to observe the drug washout restrictions
* Having been on other clinical drug/device studies in the last 30 days prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC[0-6h]) of Post-Dose FEV1 Percentage Change (∆%FEV1) from the Same-Day Pre-Dose Baseline | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. Area under the curve (AUC), from baseline to 6 hours post-dose, for the treatment period is calculated using the trapezoidal rule. Statistical analysis is performed using a one-sided t-test.

SECONDARY OUTCOMES:
Area Under the Curve (AUC[0-6h]) of Placebo Adjusted Post-Dose FEV1 Percentage Change (∆∆%FEV1) from the Same-Day Pre-Dose Baseline | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. ∆∆FEV1% for the study visit is calculated by subtracting the mean ∆%FEV1 for subjects in a randomized treatment arm from their ∆%FEV1. Area under the curve (AUC), from baseline to 6 hours post-dose, for the study visit is calculated using the trapezoidal rule.
Area Under the Curve (AUC[0-6h]) of Post-Dose FEV1 Volume Changes (∆FEV1) from the Same-Day Pre-Dose Baseline | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. Area under the curve (AUC), from baseline to 6 hours post-dose, for the treatment period is calculated using the trapezoidal rule.
Time to Onset of Bronchodilator Effect (t[onset]) | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. t[onset] is the point where post-dose ∆%FEV1 first reaches ≥ 12% over the pre-dose baseline. Determined by linear interpolation.
Peak Bronchodilator Response (F[max]) | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. F[max] is the maximum post-dose ∆%FEV1.
Time to Peak ∆FEV1 Effect (t[max]) | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. The time to peak ∆FEV1 effect, t[max], is defined as the time of F[max].
Area Under the Curve (AUC[0-6h]) of Post-Dose FEV1 in Volume from the Same-Day Pre-Dose Baseline | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. Area under the curve (AUC), from baseline to 6 hours post-dose, for the treatment period is calculated using the trapezoidal rule.
F[max] of Post-Dose FEV1 in Volume | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. F[max] of post-dose FEV1 in volume is the maximum post-dose FEV1.
Efficacy Duration-1 | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. Efficacy Duration-1 is total duration of bronchodilator effects when ∆%FEV1 is ≥ 12% above the baseline.
Efficacy Duration-2 | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. Efficacy Duration-2 is total duration of bronchodilator effects when ∆FEV1 is ≥ 200 mL above the baseline.
Efficacy Duration-3 | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. Efficacy Duration-3 is total duration of bronchodilator effects when ∆FEV1 is ≥ 100 mL above the baseline.
Bronchodilator Response | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. Subjects that demonstrate a ≥ 12% increase for ∆%FEV1 will be classified as having a bronchodilator response.
Dose Response Curve | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  The forced expiratory volume in the 1st second (FEV1) is measured with a clinically accepted model of spirometer. Subjects perform a pre-dose baseline FEV1 prior to dosing and perform subsequent FEV1 tests at 5, 15 and 30 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours after dosing during each treatment period. The dose response curve is the AUC[0-6h] of ∆%FEV1 versus study drug dosage.

OTHER OUTCOMES:
Systolic and Diastolic Blood Pressure (SBP/DBP) at Screening | Within 30 minutes prior to reversibility dosing (baseline) and 30 minutes post-reversibility dosing
  Subjects have their vital signs, i.e., blood pressure and heart rate, measured prior to reversibility dosing and 30 minutes after dosing during the Screening Visit.
Systolic and Diastolic Blood Pressure (SBP/DBP) | Within 1 hour prior to dosing (baseline) to 6 hours post-dose
  Subjects have their vital signs, i.e., blood pressure and heart rate, measured prior to dosing and at 15 and 30 minutes and 1, 1.5, 2, and 6 hours post-dose during each treatment period.
Heart Rate (HR) at Screening | Within 30 minutes prior to reversibility dosing (baseline) and 30 minutes post-reversibility dosing
  Subjects have their vital signs, i.e., blood pressure and heart rate, measured prior to reversibility dosing and 30 minutes after dosing during the Screening Visit.
Heart Rate (HR) | Within 1 hour prior to dosing (baseline) to 6 hours post-dose
  Subjects have their vital signs, i.e., blood pressure and heart rate, measured prior to dosing and at 15 and 30 minutes and 1, 1.5, 2, and 6 hours post-dose during each treatment period.
12-Lead ECG QT/QTc Intervals at Screening | Within 1 hour prior to reversibility dosing
  12-Lead ECGs are performed to measure QT and QTc intervals prior to reversibility dosing during the Screening Visit.
12-Lead ECG QT/QTc Intervals | Within 1 hour prior to dosing (baseline) to 6 hours post-dose
  12-Lead ECGs are performed to measure QT and QTc intervals prior to dosing and at 30 minutes and 1, 2, and 6 hours post-dose during each treatment period.
Number of Subjects with Incidents of Asthma Exacerbation | Participants will be followed for the duration of the study, an expected average of 3 weeks
  An asthma exacerbation incident is defined as significant worsening of clinical symptoms that cannot be adequately relieved by the rescue medication, or significant deterioration of FEV1 tests combined with clinical symptoms. Investigators monitor worsening of asthma symptoms during the treatment period and determine if subjects had experienced an asthma exacerbation.
Number of Subjects that Used Rescue Drug | Within 30 minutes prior to dosing (baseline) to 6 hours post-dose
  Rescue medication may be used to control worsening or exacerbations of asthma symptoms during the study visits when necessary, as determined by the investigator.
Complete Blood Count (CBC) at Screening | Within 1 hour after reversibility dosing
  A CBC is performed as part of the subject safety evaluations with differentials including: red blood cell (RBC), hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), and white blood cell types (WBC).
Complete Blood Count (CBC) at End-of-Study | 120 minutes post-dose at Visit 5 (within 57 days after Visit 1)
  A CBC is performed as part of the subject safety evaluations with differentials including: red blood cell (RBC), hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), and white blood cell types (WBC).
Comprehensive Metabolic Panel (CMP) at Screening | Within 1 hour after reversibility dosing
  A CMP is performed as part of the subject safety evaluations looking at levels for the following: total protein (albumin/globulin), sodium, chloride, potassium, glucose, calcium, carbon dioxide (CO2), blood urea nitrogen (BUN), creatinine, alkaline phosphate (ALP), alanine transaminase (ALT), aspartate transaminase (AST), and bilirubin.
Comprehensive Metabolic Panel (CMP) at End-of-Study | 120 minutes post-dose at Visit 5 (within 57 days after Visit 1)
  A CMP is performed as part of the subject safety evaluations looking at levels for the following: total protein (albumin/globulin), sodium, chloride, potassium, glucose, calcium, carbon dioxide (CO2), blood urea nitrogen (BUN), creatinine, alkaline phosphate (ALP), alanine transaminase (ALT), aspartate transaminase (AST), and bilirubin.
Urinalysis at Screening | Within 1 hour after reversibility dosing
  Routine and microscopic urinalysis is performed as part of the subject safety evaluations to measure urine pH and specific gravity.
Urinalysis at End-of-Study | 120 minutes post-dose at Visit 5 (within 57 days after Visit 1)
  Routine and microscopic urinalysis is performed as part of the subject safety evaluations to measure urine pH and specific gravity.
Incidents of Pregnancy at Screening | Within 1 hour prior to reversibility dosing
  A urinary pregnancy test was performed for women of child-bearing potential as a part of the Screening Visit evaluations to determine the eligibility of the subject for the study.
Incidents of Pregnancy at End-of-Study | At or after 120 minutes post-dose at Visit 5 (within 57 days after Visit 1)
  A urinary pregnancy test was performed for women of child-bearing potential as a part of the End-of-Study safety evaluations to determine if a pregnancy had occurred during the study.
Concomitant Medication Usage | Participants will be followed for the duration of the study, an expected average of 3 weeks
  Concomitant medications used by subjects throughout the duration of the study, from 30 days prior to Screening to End-of-Study evaluations, are recorded by the investigators. The total number of times a specific concomitant medication is used during the study is summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Safety Monitor, Study Director — Amphastar Pharmeceuticals, Inc.
Locations (4):
- United States (4):
  - Amphastar Site 0001, San Jose, California
  - Amphastar Site 0025, Medford, Oregon
  - Amphastar Site 0030, New Braunfels, Texas
  - Amphastar Site 0032, San Antonio, Texas

REFERENCES:
- [Background] Lipworth BJ, Clark DJ. Lung delivery of salbutamol given by breath activated pressurized aerosol and dry powder inhaler devices. Pulm Pharmacol Ther. 1997 Aug;10(4):211-4. doi: 10.1006/pupt.1997.0093. PMID 9695144
- [Background] Ahrens RC. The role of the MDI and DPI in pediatric patients: "Children are not just miniature adults". Respir Care. 2005 Oct;50(10):1323-8; discussion 1328-30. PMID 16185368
- [Background] Goldstein DA, Tan YK, Soldin SJ. Pharmacokinetics and absolute bioavailability of salbutamol in healthy adult volunteers. Eur J Clin Pharmacol. 1987;32(6):631-4. doi: 10.1007/BF02456001. PMID 3653233
- [Background] Hindle M, Newton DA, Chrystyn H. Dry powder inhalers are bioequivalent to metered-dose inhalers. A study using a new urinary albuterol (salbutamol) assay technique. Chest. 1995 Mar;107(3):629-33. doi: 10.1378/chest.107.3.629. PMID 7874928
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Crapo RO, Morris AH, Gardner RM. Reference spirometric values using techniques and equipment that meet ATS recommendations. Am Rev Respir Dis. 1981 Jun;123(6):659-64. doi: 10.1164/arrd.1981.123.6.659. PMID 7271065
- [Background] Crapo RO, Morris AH, Clayton PD, Nixon CR. Lung volumes in healthy nonsmoking adults. Bull Eur Physiopathol Respir. 1982 May-Jun;18(3):419-25. PMID 7074238